CLINICAL TRIAL: NCT00004374
Title: Study of Systemic Amyloidosis Presentation and Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Indiana University School of Medicine (Other)
Other Study IDs: NCRR-M01RR00750-0062; IUSM-831215
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Amyloidosis
Keywords: amyloidosis; arthritis & connective tissue diseases; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Amyloidosis; Arthritis; Connective Tissue Diseases; Genetic Diseases, Inborn; Rare Diseases

SUMMARY:
OBJECTIVES: I. Analyze prospectively the course of amyloid deposition in patients with primary, secondary, myeloma-associated, and hereditary amyloidosis.

II. Determine abnormalities of humoral and delayed-type hypersensitivity in these patients.

III. Identify prognostic factors in hereditary amyloidosis and develop tests for genetic defects associated with systemic amyloidosis.

IV. Diagnose familial amyloidotic polyneuropathy (FAP) prior to symptom onset. V. Validate the correlation of low serum prealbumin and retinol binding protein levels with amyloidosis in patients with FAP.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive a comprehensive evaluation with an emphasis on identifying prognostic and diagnostic factors. Assessments include gastrointestinal, renal, hematologic, dermatologic, cardiac, and serologic studies. Immunologic studies include antinuclear antibody, latex fixation, and serum and urine electrophoresis.

Genetic trees are constructed using detailed family history data; blood and urine samples are routinely collected from relatives. Family members of patients with familial amyloidotic polyneuropathy type II (Indiana type) undergo a flexor retinaculum biopsy of the wrist.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Systemic amyloidosis, i.e.: Primary, myeloma associated Secondary, e.g., associated with the following conditions: Rheumatoid arthritis Inflammatory bowel disease

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1979-01

CONTACTS AND LOCATIONS:
Overall Officials: Merrill D. Benson, Study Chair — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States